CLINICAL TRIAL: NCT04039243
Title: Addressing Anxiety in 2-Year-Olds: A Pilot Screening and Intervention Study
Brief Title: Addressing Anxiety in 2-3-Year-Olds: A Pilot Intervention Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dina R. Hirshfeld-Becker, Co-Director, MGH Child CBT Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P000376
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorder of Childhood; Fear; Shyness
Keywords: Anxiety disorders; Toddlers; Preschoolers; Cognitive-behavioral therapy
MeSH Terms: conditions — Shyness; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Treatment (Experimental): Up to 12 sessions of Parent-Child CBT using an adaptation of the Being Brave protocol
  Interventions: Behavioral: Being Brave
- Parent Education (Active Comparator): Parents receive educational materials about how to help young children overcome shyness and anxiety
  Interventions: Other: Parent Education
- Monitoring (No Intervention)

INTERVENTIONS:
Behavioral: Being Brave — Up to 12 weekly sessions
  Arms: Active Treatment
Other: Parent Education — Parents receive educational materials about helping children overcome shyness and fear
  Arms: Parent Education

SUMMARY:
The purpose of this study is to test the feasibility and efficacy of intervening with 2-year-old children with elevated temperamental Fear and/or Shyness or 3-year-old children with elevated anxiety and their parents, using a parent-child Cognitive Behavioral Therapy (CBT) protocol to reduce anxiety disorders and maintain reduced anxiety at one-year follow-up. Before the COVID-19 pandemic, study visits and treatment sessions were conducted in office. Now all visits and treatment sessions are conducted remotely.

ELIGIBILITY:
Inclusion Criteria:

* The child scores >1 Standard Deviation (SD) above reported means for the Fear or Shyness scales on the Early Childhood Behavior Questionnaire (ECBQ) (if child is 21-35 months) or the child scores >1SD above reported means for the Total Anxiety, Generalized Anxiety, Social Anxiety, Physical Injury Fears, or Separation Anxiety scales on the Preschool Anxiety Scale (PAS) (if child is 36-47 months) as completed by a parent
* The parents are able to speak, understand, and read English
* The child must have a working knowledge of English.

Exclusion Criteria:

* Autism Spectrum Disorder (ASD) or global developmental delay in the child
* The child has disruptive behavior so severe as to interfere with participation in intervention sessions
* The child has a different primary disorder for which CBT for anxiety is inappropriate (e.g. severe depression, depression in the mother, significant medical disorder).

Ages: 21 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-09-27 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Response Rate (proportion of participants rated as 1 or 2 on Clinical Global Impression of Anxiety-Improvement Measure (CGI-I) | Baseline to four-month follow-up
  The CGI-I is a 7-point scale from 1 (Very Much Improved) to 7 (Very Much Worse). It will be rated by a clinician interviewer blind to treatment condition
CGI-Severity Ratings | Compared between groups at 4- and 8-month FU

CONTACTS AND LOCATIONS:
Overall Officials: Dina Hirshfeld-Becker, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States